CLINICAL TRIAL: NCT02735681
Title: Effect of Meibomian Gland Probing on Ocular Surface in Ocular Rosacea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trouble recruiting
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205144
Record Dates: First submitted 2016-03-29; First posted 2016-04-13 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probing Treatment Right Eye (Active Comparator): Meibomian gland will be performed on the right upper eye lid of each participant.
  Interventions: Procedure: meibomian gland probing
- Fellow Eye (Left) Untreated (Placebo Comparator): The fellow eye (left) will be used at the untreated control
  Interventions: Procedure: Left eye Meibomian Gland Probing Control Group

INTERVENTIONS:
Procedure: meibomian gland probing — Investigator will do baseline (OSDI) questionnaires prior to probing as well as at 1 week (at home), 1 month, 3months, and 6 months at office visits.
  Arms: Probing Treatment Right Eye
Procedure: Left eye Meibomian Gland Probing Control Group — There will be no probing in the left eye. This will be used as a control for the right eye.
  Arms: Fellow Eye (Left) Untreated

SUMMARY:
Meibomian glands (MG) are modified sebaceous glands associated with the tarsus (collagenous structural component) of the upper and lower eyelids. Meibomian glands produce lipid-based secretions which are an integral and stabilizing part of the tear film. In blepharitis and ocular rosacea (two known causes of obstructive meibomian gland dysfunction (o-MGD), inflammation of the lid margins causes blockage of the meibomian gland orifices, changes in glandular secretions, and dropout of the glands themselves. This limits the production, secretion, and quality of meibum. With less oil in the tear film, the aqueous portion of tears is not stable and evaporates quickly which leads to dry eye.

DETAILED DESCRIPTION:
Meibomian gland probing is a relatively new, safe, and effective technique for treating obstructive meibomian gland dysfunction (o-MGD). It involves topical anesthesia of the eyelid margins and insertion of a 2 mm or 4 mm sterile, beveled, solid stainless steel probe at the slit lamp. Meibomian gland probing has been reported to alleviate symptoms (lid tenderness / lid margin congestion) of o-MGD (Maskin, 2010). It has also been shown to improve meibum lipid levels, viscosity, and tear breakup time (Nakayama, Kawashima, Kaido, Arita, & Tsubota, 2015). Though probing has been investigated in a few small studies of o-MGD, only one small study of 10 participants has investigated meibomian gland probing in ocular rosacea (Wladis, 2012). This study showed improvement in ocular surface disease index (OSDI, a standardized questionnaire assessing dry eye) but did not show objective improvement by way of examination findings or analysis of meibum (Wladis, 2012).

In our study, Investigators intend to further investigate meibomian gland probing in participants with diagnosed ocular rosacea. Investigators hypothesize that after probing of one eye, Investigators will note improvements in participants symptoms as reflected in improvement in OSDI scores, Reductions in Inflamma-Dry measures (measure of matrix metalloproteinase (MMP-9), an inflammatory marker elevated in tears of participants with dry eye), decreased tear fluid osmolarity, decreased meibum viscosity on expression . Objective improvement in lid margin disease (noting collarettes, pitting, telangiectasia of lid margins, thickening / irregularity of lid margins, lid margin tenderness; improvement in tear break up time (TBUT); and improvement in corneal fluorescein / lissamine green staining).

ELIGIBILITY:
Inclusion Criteria:

• Diagnosed Ocular Rosacea +/- Facial Rosacea

Exclusion Criteria:

* Prior meibomian gland probing
* Prior treatment with Lipiflow
* Cicatricial Disease
* Sjogren's Syndrome
* Prior radiation therapy to face / head
* Allergy to lissamine green and fluorescein

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Improvements in participants symptoms as reflected in improvement in Ocular Surface Disease Index (OSDI) scores | Up to 6 months
  The OSDI is assessed on a scale of 0 and 100, with higher scores representing greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Sunali Goyal, MD, Principal Investigator — University of Arkansas; Joshua Hardin, MD, Principal Investigator — University of Arkansas
Locations (1):
- Jones Eye Institute, UAMS, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No